CLINICAL TRIAL: NCT03176173
Title: Radical-Dose Image Guided Radiation Therapy in Treating Patients With Metastatic Non-small Cell Lung Cancer Undergoing Immunotherapy
Brief Title: Radical RADiotherapy and Immunotherapy for Metastatic CAncer of the Lung (RRADICAL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Michael Francis Gensheimer, Clinical Associate Professor, Radiation Oncology - Radiation Therapy, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-40088; NCI-2017-00952 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0088 (Other: OnCore)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-08

CONDITIONS: Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Image-Guided; Immunotherapy; Biological Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunotherapy plus Image-guided Radiation Therapy (Experimental): Patients undergo radical-dose image guided radiation therapy daily for up to 10 days (within 2 weeks) while continuing their prior treatment with the treating physician's choice of regular medical care immunotherapy.
  Interventions: Radiation: Image-guided Radiation Therapy; Drug: Immunotherapy (physician's choice for standard of care immunotherapy)
- Immunotherapy Alone (Regular Medical Care) (Active Comparator): Patients who decline to undergo radiation therapy will continue their prior treatment with the treating physician's choice of regular medical care immunotherapy.
  Interventions: Drug: Immunotherapy (physician's choice for standard of care immunotherapy)

INTERVENTIONS:
Radiation: Image-guided Radiation Therapy — Ablative treatment as 50 Gy in 5 or 10 fractions.
  Non-ablative treatment as 27 Gy in 3 fractions, or 40 Gy in 10 fractions.
  Other Names: IGRT
  Arms: Immunotherapy plus Image-guided Radiation Therapy
Drug: Immunotherapy (physician's choice for standard of care immunotherapy) — Continue regular medical care immunotherapy. Other than being an anti-PD-1 or anti-PD-L1 immunotherapy, the agent, dose, and schedule is not specified by protocol.
  Other Names: biologic therapy

SUMMARY:
This phase II trial studies how well radical-dose image guided radiation therapy works in treating patients with non-small cell lung cancer that has spread to other places in the body who are undergoing immunotherapy. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radical-dose image guided radiation therapy to patients with non-small cell lung cancer may help to improve response to immunotherapy anti-cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if progression-free survival at 24 weeks with this treatment combination is improved compared to historical controls who received immunotherapy without radiation therapy.

SECONDARY OBJECTIVES:

I. Assess acute (0-6 months) and late (> 6 months) grade 3-5 toxicity. II. Assess overall survival. III. Correlate circulating tumor deoxyribonucleic acid (DNA) (ratio of post-radiation therapy [RT] to pre-RT level) with radiographic response.

IV. Correlate immune markers in peripheral blood with radiographic response.

TERTIARY OBJECTIVES:

I. Analyze progression-free survival with immune-related response criteria. II. Measure time to discontinuation of study immunotherapy agent. III. Assess patterns of progression.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients undergo radical-dose image guided radiation therapy daily for up to 10 days (within 2 weeks) while undergoing standard of care immunotherapy.

Arm II: Patients who decline to undergo radiation therapy receive standard of care immunotherapy.

After completion of study treatment, patients are followed up at 30 days and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Has stage IV non-small cell lung cancer, or initially stage I-III disease with distant metastatic recurrence
2. Age ≥ 18
3. Has been receiving anti-PD-1 or anti-PD-L1 immunotherapy for at least four weeks (refer to section 4.2.1)
4. Has had restaging imaging after initiation of immunotherapy, at least 4 weeks after pre-immunotherapy baseline imaging. CT or PET/CT of at least chest/upper abdomen must be performed within 4 weeks prior to registration. For patients with history of brain metastases, brain MRI or CT is required within 4 weeks of registration; for other patients brain MRI or CT is required within 12 weeks of registration. Diagnostic PET/CT performed as part of radiation simulation can be used as the restaging imaging.
5. Most recent imaging shows measurable disease as defined by RECIST 1.1
6. Evaluation by a Stanford medical oncologist must show:

   1. The patient is expected to continue on immunotherapy for at least three more months
   2. Imaging must show response, stable disease, or modest progression
   3. If there is modest progression, the patient must be clinically stable in terms of performance status and overall disease-related symptoms
7. Has at least one extracranial tumor safely treatable with radical-dose radiation therapy and that has not been previously treated with radiation
8. ECOG performance status 0-2
9. Has the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Untreated brain metastases, if not planned to be treated in this course of radiation therapy
* Pregnancy or women of childbearing potential not willing/able to use contraception during protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gensheimer, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although the 'Immunotherapy Alone (Regular Medical Care)' arm was included in the study design, no participants were enrolled or assigned to this arm
Groups:
- Immunotherapy Plus Image-guided Radiation Therapy: Patients undergo radical-dose image guided radiation therapy daily for up to 10 days (within 2 weeks) while continuing their prior treatment with the treating physician's choice of regular medical care immunotherapy.
  Image-guided Radiation Therapy: Ablative treatment as 50 Gy in 5 or 10 fractions.
  Non-ablative treatment as 27 Gy in 3 fractions, or 40 Gy in 10 fractions.
  Immunotherapy (physician's choice for standard of care immunotherapy): Continue regular medical care immunotherapy. Other than being an anti-PD-1 or anti-PD-L1 immunotherapy, the agent, dose, and schedule is not specified by protocol.
Period: Overall Study
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy | Immunotherapy Alone (Regular Medical Care)
Started | 45 | 0
Completed | 44 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only participants were enrolled in Arm 1 (Immunotherapy plus Image-guided Radiation Therapy); therefore, no baseline data are available for Arm 2 (Immunotherapy Alone).
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy | Immunotherapy Alone (Regular Medical Care) | Total
Number analyzed (Participants) | 44 | 0 | 44
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2 |  | 2
  40-49 years | 3 |  | 3
  50-59 years | 4 |  | 4
  60-69 years | 10 |  | 10
  70-79 years | 18 |  | 18
  80-89 years | 7 |  | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 |  | 19
  Male | 25 |  | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 43 |  | 43
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 15 |  | 15
  Native Hawaiian or Other Pacific Islander | 2 |  | 2
  Black or African American | 0 |  | 0
  White | 26 |  | 26
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 44 |  | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Defined as percentage of participants without disease progression or death at 24 weeks from date of study entry, assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): ≥30% decrease in the sum of the longest diameter of target lesions
  Overall Response (OR): CR + PR
Time Frame: 24 weeks from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 43
Participants | 26
Statistical Analysis 1: Comparison: Immunotherapy Plus Image-guided Radiation Therapy; Test type: Superiority; p = 0.0007, Exact binomial test

2. Secondary Outcome: Change in Circulating Tumor Deoxyribonucleic Acid Levels as Measured Using CAncer Personalized Profiling by Deep Sequencing
Description: Will correlate with radiographic response. Plasma biomarkers (e.g. cell free deoxyribonucleic acid level) will be summarized using medians and interquartile ranges; changes in biomarkers will be assessed using the Wilcoxon signed rank test. Correlation of biomarkers with radiographic response will be evaluated using a Wilcoxon rank sum test on patients with and without the event of interest. If feasible, these analyses will be supplemented by more formal analyses with the Cox model.
Time Frame: Baseline (pre-treatment)
Population: Blood samples were collected for this outcome measure, however, no laboratory analysis was conducted due to lack of funding. No future analyses are planned.
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Immune Marker Levels as Measured From Peripheral Blood Using Flow Cytometry Performed by the Human Immune Monitoring Core at Stanford University
Description: Change in immune marker levels was measured using flow cytometry performed by the Human Immune Monitoring Core at Stanford University. These changes will correlate with radiographic response.
Time Frame: Pre-radiation (up to 14 days before RT) and post-radiation (up to 14 days after completion of RT)
Population: Peripheral blood samples were collected at the pre-specified time points, but immune marker levels were not analyzed due to lack of funding for laboratory processing. No future analyses are planned.
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Acute (0-6 Months) and Late (> 6 Months) Grade 3-5 Toxicity
Description: This outcome measured the number of participants who experienced Grade 3-5 acute (0-6 months) and late (>6 months) toxicities, assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4, through up to 4 years after study entry.
Time Frame: Up to 4 years after study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 44
Participants | 4

5. Secondary Outcome: Overall Survival
Description: The electronic medical record was monitored for patient deaths.
Time Frame: Time from study entry to death, assessed up to 4 years after study entry
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 44
months | 27.4 [20.37 to NA] — The upper bound of the 95% confidence interval could not be estimated due to an insufficient number of events at later time points.

6. Other Pre Specified Outcome: Number of Participants With Tumor Response (Including Abscopal Responses)
Description: Number of participants who experienced a tumor response, including abscopal responses, following image-guided radiation therapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 44
Participants | 26

7. Other Pre Specified Outcome: Progression Free Survival
Description: Evaluated with immune-related Response Criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Pre-radiation (up to 14 days before RT) and post-radiation (up to 14 days after completion of RT)
Population: Imaging data were collected for assessment of progression-free survival using immune-related response criteria (iRRC); however, these data were not analyzed because the outcome was deemed not scientifically relevant at the time of final analysis. No future analyses are planned.
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Time to Discontinuation of Study Immunotherapy Agent
Description: Time to discontinuation of study immunotherapy agent was measured.
Time Frame: Up to 4 years
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
Number analyzed (Participants) | 44
Months | 6.1 [2.7 to 12.8]

ADVERSE EVENTS:
Time Frame: 4 years
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Immunotherapy Plus Image-guided Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/44
Serious Adverse Events (participants affected / at risk) | 6/44
Other Adverse Events (participants affected / at risk) | 32/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy Plus Image-guided Radiation Therapy (N=44)
Other - Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy Plus Image-guided Radiation Therapy (N=44)
Fatigue (General disorders) | 25 (36)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Other - Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (22)
Anorexia (Metabolism and nutrition disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24)
Esophagitis (Gastrointestinal disorders) | 8 (9)
Dermatitis radiation (Injury, poisoning and procedural complications) | 7 (8)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Toothache (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Several pre-specified biomarker and imaging outcomes were not analyzed due to lack of funding for laboratory processing or because analyses were deemed not scientifically relevant at the time of final review. No future analyses are planned for these measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT03176173/Prot_000.pdf